CLINICAL TRIAL: NCT05616208
Title: Phase 1 Treatment Study to Assess Safety and Proof of Concept to Assess Potential Efficacy of the Implanted Internal Anal Sphincter BioSphincterTM Bioengineered From Autologous Cells to Treat Patients With Severe Passive Fecal Incontinence
Brief Title: Implantation of BioSphincter TM for Treatment of Severe Passive Fecal Incontinence
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cellf Bio LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2022-10-31; First posted 2022-11-15 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Fecal Incontinence
Keywords: fecal incontinence; accidental bowel leakage; fecal urgency
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: This is a non-randomized, single group treatment study with a single arm and is not subject or investigator masked or blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Implantation (Experimental): This is a non-randomized, single group treatment study with a single arm and is not subject or investigator masked or blinded. BioSphincters will be implanted in every study subject.
  Interventions: Biological: Bioengineered Internal Anal Sphincter

INTERVENTIONS:
Biological: Bioengineered Internal Anal Sphincter — Autologous Bioengineered Internal Anal Sphincter
  Other Names: BioSphincter(TM)

SUMMARY:
This is first-in-human prospective Phase I study of the immediate and long-term safety of an implanted internal anal sphincter (IAS) bioengineered from autologous cells to treat subjects with severe passive FI who have failed standard treatments.

DETAILED DESCRIPTION:
This is a two-center first-in-human prospective Phase I study of the immediate and long-term safety of an implanted internal anal sphincter (IAS) bioengineered from autologous cells to treat subjects with severe passive FI who have failed standard treatments. The data will be analyzed to assess the safety of the treatment and the potential initial efficacy of the implanted BioSphincter(TM) in decreasing the number of episodes of incontinence in subjects with severe FI.

After being informed of the risks, informed consent patients will undergo a biopsy procedure to collect tissue samples and will then undergo an implantation surgery of the bioengineered BioSphincter(TM). Patients will be followed for 36 months, post implantation.

ELIGIBILITY:
Inclusion Criteria

Patients are eligible to be included in the study only if all of the following criteria apply:

1. Males and females aged 18 years old and over at the time of signing the IRB approved informed consent.
2. Have the ability to understand the requirements of the study and are willing to comply with all study procedures.
3. In the opinion of the investigator, able to participate in the study.
4. Experience four or more FI episodes per 2-week period for the past 12 months. For purposes of this study, FI is defined as the loss of control sufficient to have stool in the subject's undergarments or require the changing of the undergarments. FI does not include the presence of a minimal amount of fecal material on the subject's undergarments and does not require the changing of the undergarments.
5. Failed standard medical and surgical therapies for FI as defined below:

   1. Failure of standard medical therapy is defined as

      * Bulking agents such as Citrucel or Metamucil fail to decrease the frequency of FI episodes to 4 or fewer episodes per two-week period after 4 weeks of treatment. Treatment failure is defined as a lack of response to the intervention after 4 weeks of treatment. Upon initiation of fiber, patients should see a change in stool consistency within 24-48 hours. Additional time for fiber treatment is needed to titrate the dose to optimize stool consistency and minimize side effects of bloating and increased flatus. Four weeks allows time to change stool consistency and measure changes in FI with a stable fiber regimen.
      * Antidiarrheal agents such as Imodium or Lomotil may decrease FI or produce constipation but fail to decrease the frequency of FI episodes to 4 or fewer episodes per two-week period after 4 weeks of treatment. Treatment failure is defined as a lack of response to the intervention after 4 weeks of treatment. Upon initiation of Imodium or Lomotil, the patient should see a change in stool frequency within 24-48 hours. Additional time on Imodium/Lomotil treatment is needed to titrate the dose to optimize stool frequency and minimize side effects of bloating. Four weeks allows time to change stool frequency and measure changes in FI on a stable Imodium/Lomotil regimen.
      * Failure of biofeedback training to reduce the frequency of FI episodes to 4 or fewer episodes per two-week period after 4 weeks of treatment. Treatment failure is defined as a lack of response to the intervention after 3 months of treatment. Three months of physical therapy is needed to allow strengthening of pelvic floor musculature and improvement in pelvic floor coordination.
   2. Failure of standard surgical therapy is defined as

      * Sacral nerve stimulation (SNS) fails to decrease the frequency of FI episodes to 4 or fewer episodes per two-week period after 2 months or more of treatment. SNS requires a two week period for two surgeries, trial implantation and then permanent implantation. During the two week period, patients can see a change in FI symptoms secondary to SNS implantation that informs the decision to proceed with permanent implantation. After permanent implantation, the settings of the SNS can be manipulated to optimize fecal control and minimize patient side effects. Two months allows time for the two surgeries to occur and SNS setting changes to ensure optimization of FI. Failure of SNS treatment will also include patients who have SNS explantation due to complications or side effects. Finally, SNS failure will also include patients who fail test stimulation and do not undergo chronic implantation. Patients can be considered to have SNS failure if after informed consent for the procedure, they elect to not undergo SNS trial or implantation.
      * Sphincteroplasty failure will have occurred if the FI episode frequency is four or more episodes per two-week period, 12 months or more after surgical repair. After sphincteroplasty, patients may initially see an improvement in FI. However, over time, there has been a measured degradation in response to this surgical despite intact sphincter repair. Therefore, after 12 months, if a patient has undergone sphincteroplasty but fails to have improvement in FI, OR redevelops FI after initial improvement in FI, the patient will be eligible for potential trial enrollment.
   3. Patients with severe passive fecal incontinence are eligible for the trial if they have failed all medical and surgical therapy for fecal incontinence and are being considered for a colostomy.
6. Anorectal manometry (ARM) testing history of ARM while at the discretion of the Physician/Surgeon. ARM must show low IAS pressure and presence of the Recto Anal Inhibitory Reflex (RAIR). Low IAS pressure is defined as ≤ 60 mmHg during the anorectal motility exam performed with a high-resolution catheter. Normal IAS pressure range is > 60 mm Hg.
7. Pre-surgery, vital signs must be within the following parameters: SBP (mmHg) >100 or < 140; DBP (mmHg) >60 or <90; HR >60 or <100 bpm; afebrile, RR< 20 or >12 bpm; Pulse ox >95% on room air.
8. Women of childbearing potential must use acceptable contraceptives during this study. Acceptable contraceptives include oral contraceptives and IUDs. Females of childbearing potential will have a urine pregnancy test on the day of trial enrollment.
9. Women not using hormonal contraception or hormonal replacement therapy (HRT) must have confirmation of a postmenopausal state. A high follicle stimulating hormone (>40 IU/L) level in the postmenopausal range may be used; however, in the absence of 12 months of amenorrhea, confirmation with more than one FSH measurement is required.
10. Men of childbearing potential should use a medically accepted contraceptive during this study. Acceptable contraceptives include total abstinence and condoms + spermicide.
11. Colonoscopy performed within the past 5 years that excludes malignancy, inflammation, or infection.
12. Willingness to return for all follow-up visits through 36 months post-treatment.

Exclusion Criteria

A patient is not eligible for inclusion in the study if any of the following criteria apply:

1. Symptomatic anorectal disease including hemorrhoid disease, anal fissure, or fistula causing symptoms such as bleeding, swelling, pain, or drainage.
2. Pre-existing anorectal pain of any cause.
3. Incontinence of flatus only.
4. Chronic watery diarrhea unmanaged by medical therapy and which is the primary cause for FI.
5. Greater than 60 degrees of either external anal sphincter disruption or both (>60° IAS and EAS). Patients with severe (>60 degree) disruption of the EAS ± IAS are likely to have a component of both urge (EAS) and passive (IAS) fecal incontinence. Due to a combined etiology of FI, patients with a large EAS ± IAS disruption are unlikely to have a significant improvement in FI from BioSphincter treatment.
6. Acute or chronic anorectal infections (including proctitis, recurrent abscesses, or fistulae).
7. Presence of anorectal tumors.
8. Active proctitis.
9. Uncontrolled inflammatory bowel disease (IBD) characterized by one or more of the following: CRP 10 mg/L, fecal calprotectin > 200 mg/L, new or uncontrolled symptoms of IBD, endoscopic disease, evidence of inflammation on MR Imaging.
10. Any illness or disease requiring chemotherapy or any malignant disease within 5 years of enrollment.
11. History of organ transplantation requiring immunosuppressive medications.
12. History of a bleeding disorder diagnosed and treated by a hematologist, or patient with a diagnosed bleeding disorder currently being treated by a hematologist. If patient is on anticoagulation therapy which can be temporarily halted with permission from the prescribing provider for elective surgery, the patient will be eligible for the trial.
13. History of pelvic radiation, rectal prolapse, anorectal malformations, anorectal surgery within the previous 12 months or current colostomy..
14. Neurologic disease characterized by significant peripheral neuropathy or spinal cord dysfunction.
15. Mobility impairment requiring the use of assistive devices (e.g., wheelchair).
16. Current pregnancy, breastfeeding, or childbirth within previous 12 months.
17. History of unstable cardiac function (New York Heart Association Functional Classification III or IV).
18. History of unstable pulmonary function requiring home oxygen.
19. History of abnormal kidney function (Cr >1.5 mg/dl or on dialysis).
20. Any clinically important abnormal laboratory tests, including but not limited to:

    1. Hemoglobin <10g.
    2. ALT and AST >2 times the upper limit of normal).
    3. Bilirubin >1.5mg/dl. For criteria a, b, and c, the test can be repeated one time at the discretion of the Investigator. If this option is used, the last obtained reading will be used for determination of eligibility. Averages will not be used.
21. Active untreated gynecological or urologic infection.
22. Documented history of or positive test results for human immunodeficiency virus (HIV)-1/HIV-2 Antibodies (Abs), Hepatitis B surface Antigen (HBsAg), or Hepatitis C Antibody (HCVAb) and evidence of a chronic active infection.
23. Presence of significant comorbidities that may be an underlying cause of FI (e.g., uncontrolled diabetes (>7.5 HgA1C), severe spinal stenosis).
24. History of alcohol or substance abuse within past 12 months.
25. Concurrent participation in any other clinical investigation during the period of this investigation. Patients who have been treated with any other investigational drug or participated in any investigational study within 30 days prior to enrollment in this study.
26. Inability to participate in all necessary study activities due to physical or mental limitations.
27. Inability or unwillingness to return for all required follow-up visits.
28. Inability or unwillingness to sign informed consent.
29. Any circumstance in which the investigator deems that participation in the study is not in the subject's best interest.
30. Presence of increased surgical risk associated with jejunal or IAS biopsy (e.g., multiple previous surgeries with potential for adhesions, ventral hernia). Subjects also may be excluded during the biopsy procedure (i.e., an intraoperative exclusion) if the investigator observes any conditions that in the investigator's opinion would generate increased risk. Should this occur, biopsy will not be performed, and the subject will be classified as an intraoperative screen failure.
31. Previous history of anorectal surgery or disease which would prevent or increase the difficulty of surgical dissection of the intersphincteric space.
32. Allergy to Marcaine, epinephrine, betadine, Dermabond dressing, Prolene (polypropylene) suture, Polydioxanone suture (PDS) and Monocryl suture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events of Implanted BioSphincter IAS for patients with severe FI Who Have Failed Standard Treatment | 12-36 months
  To determine the safety of IAS cell harvest and the implanted BioSphincter IAS in subjects with severe FI. Occurrence of adverse events.
  * Occurrence, severity, duration, and relationship to study procedures.
  * The safety of all surgical and diagnostic procedures will be assessed at inpatient hospital follow-up and outpatient clinic visits at predefined intervals.
    * Biopsy: Site of IAS cell harvest will be assessed postoperatively at Days 1, 7, and 21.
    * BioSphincter implantation will be assessed postoperatively at postoperative Days 1, 3, 7, 14, 28, 42 (week 6) and 56 (week 8). Additional safety assessments will be made at medical visits on Weeks 12, 24, 36 and 48-post implantation. Final safety assessments will be made a.t the end of Years 2 and 3

SECONDARY OUTCOMES:
Initial efficacy of the implanted IAS in decreasing the number of episodes of incontinence in subjects with severe FI. | 12-48 weeks
  Change in the number of FI episodes within a two-week period of each follow-up visit (at 12, 24, 36, and 48 weeks after implantation) as recorded in subjects' bowel diaries.
Initial efficacy of the implanted IAS in decreasing the number of episodes of fecal urgency in subjects with severe FI. | 12-48 weeks
  Change in the number of episodes of fecal urgency within a two-week period of each follow-up visit (at 12, 24, 36, and 48 weeks after implantation) as recorded in subjects' bowel diaries.
Change from Baseline CCIS Score of the implanted IAS in improving quality of life | 12-48 weeks
  Change in Cleveland Clinic Incontinence Score (CCIS) as evaluated at the time of each follow-up visit (at 12, 24, 36, and 48 weeks after implantation) and compared to baseline measures. Scored from 0 to 20 (0=complete continence, 20=complete incontinence)
Change from Baseline FISI Score of the implanted IAS in improving quality of life | 12-48 weeks
  Change in Fecal Incontinence Severity Index (FISI) as evaluated at the time of each follow-up visit (at 12, 24, 36, and 48 weeks after implantation) and compared to baseline measures. 0 to 61, where the higher the score, the higher the perceived severity of the fecal incontinence.
Change from Baseline FIQOL Score of the implanted IAS in improving quality of life | 12-48 weeks
  Change in Fecal Incontinence Quality of Life Scale (FIQOL) as evaluated at the time of each follow-up visit (at 12, 24, 36, and 48 weeks after implantation) and compared to baseline measures. Scales range from 1 to 5, with 1 indicating a lower functional quality-of-life status.
Initial efficacy of the implanted IAS by conducting Anal Rectal Manometry (ARM) measuring IAS pressure to support measured clinical changes | 0-36 months
  Measure of IAS pressure (mmHg) as evaluated at 12, 24, 36, and 48 weeks and at 2 and 3 years after implantation as compared with baseline measures and control subject normal values.
Initial efficacy of the implanted IAS by conducting Anal Rectal Manometry (ARM) measuring EAS pressure to support measured clinical changes | 0-36 months
  Measure EAS pressure in mmHg as evaluated at 12, 24, 36, and 48 weeks and at 2 and 3 years after implantation as compared with baseline measures and control subject normal values.
Initial efficacy of the implanted IAS by conducting Anal Rectal Manometry (ARM) measuring sensation of balloon distention pressure to support measured clinical changes | 0-36 months
  Measure time to sensation of balloon distention (in seconds) as evaluated at 12, 24, 36, and 48 weeks and at 2 and 3 years after implantation as compared with baseline measures and control subject normal values.
Initial efficacy of the implanted IAS by conducting Anal Rectal Manometry (ARM) measuring presence of RAIR to support measured clinical changes | 0-36 months
  Measure presence or absence of RAIR as evaluated at 12, 24, 36, and 48 weeks and at 2 and 3 years after implantation as compared with baseline measures and control subject normal values.
Measure Physical characteristics of the Bioengineered Sphincter as assessed by endoscopic ultrasound (EUS) | 0-36 months
  Measure physical characteristics of the thickness ( in mm) Bioengineered Sphincter as assessed by endoscopic ultrasound at 48 weeks, 2 years and 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Bohl, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University Health Main Hospital (VCU), Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baxter NN, Rothenberger DA, Lowry AC. Measuring fecal incontinence. Dis Colon Rectum. 2003 Dec;46(12):1591-605. doi: 10.1007/BF02660762. PMID 14668583
- [Background] Bharucha AE, Fletcher JG, Seide B, Riederer SJ, Zinsmeister AR. Phenotypic variation in functional disorders of defecation. Gastroenterology. 2005 May;128(5):1199-210. doi: 10.1053/j.gastro.2005.03.021. PMID 15887104
- [Background] Cleveland Clinic Incontinence Score. Vol. 0, 2021, p. 1993.
- [Background] Engel AF, Kamm MA, Bartram CI, Nicholls RJ. Relationship of symptoms in faecal incontinence to specific sphincter abnormalities. Int J Colorectal Dis. 1995;10(3):152-5. doi: 10.1007/BF00298538. PMID 7561433
- [Background] Farouk R, Duthie GS, Pryde A, McGregor AB, Bartolo DC. Internal anal sphincter dysfunction in neurogenic faecal incontinence. Br J Surg. 1993 Feb;80(2):259-61. doi: 10.1002/bjs.1800800250. PMID 8443675
- [Background] Fecal Incontinence Quality of Life Scale (FIQOL). 2021.
- [Background] Fecal Incontinence Severity Index ( FISI ). 2021.
- [Background] Goode PS, Burgio KL, Halli AD, Jones RW, Richter HE, Redden DT, Baker PS, Allman RM. Prevalence and correlates of fecal incontinence in community-dwelling older adults. J Am Geriatr Soc. 2005 Apr;53(4):629-35. doi: 10.1111/j.1532-5415.2005.53211.x. PMID 15817009
- [Background] Huebner M, Margulies RU, Fenner DE, Ashton-Miller JA, Bitar KN, DeLancey JO. Age effects on internal anal sphincter thickness and diameter in nulliparous females. Dis Colon Rectum. 2007 Sep;50(9):1405-11. doi: 10.1007/s10350-006-0877-7. PMID 17665265
- [Background] Jorge JM, Wexner SD. Etiology and management of fecal incontinence. Dis Colon Rectum. 1993 Jan;36(1):77-97. doi: 10.1007/BF02050307. PMID 8416784
- [Background] Luo C, Samaranayake CB, Plank LD, Bissett IP. Systematic review on the efficacy and safety of injectable bulking agents for passive faecal incontinence. Colorectal Dis. 2010 Apr;12(4):296-303. doi: 10.1111/j.1463-1318.2009.01828.x. Epub 2009 Mar 6. PMID 19320664
- [Background] Maeda Y, Laurberg S, Norton C. Perianal injectable bulking agents as treatment for faecal incontinence in adults. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD007959. doi: 10.1002/14651858.CD007959.pub3. PMID 23450581
- [Background] Norton C, Cody JD. Biofeedback and/or sphincter exercises for the treatment of faecal incontinence in adults. Cochrane Database Syst Rev. 2012 Jul 11;2012(7):CD002111. doi: 10.1002/14651858.CD002111.pub3. PMID 22786479
- [Background] Omar MI, Alexander CE. Drug treatment for faecal incontinence in adults. Cochrane Database Syst Rev. 2013 Jun 11;2013(6):CD002116. doi: 10.1002/14651858.CD002116.pub2. PMID 23757096
- [Background] Rao SS. Pathophysiology of adult fecal incontinence. Gastroenterology. 2004 Jan;126(1 Suppl 1):S14-22. doi: 10.1053/j.gastro.2003.10.013. PMID 14978634
- [Background] Rockwood TH, Church JM, Fleshman JW, Kane RL, Mavrantonis C, Thorson AG, Wexner SD, Bliss D, Lowry AC. Fecal Incontinence Quality of Life Scale: quality of life instrument for patients with fecal incontinence. Dis Colon Rectum. 2000 Jan;43(1):9-16; discussion 16-7. doi: 10.1007/BF02237236. PMID 10813117
- [Background] Sangwan YP, Coller JA, Schoetz DJ, Roberts PL, Murray JJ. Spectrum of abnormal rectoanal reflex patterns in patients with fecal incontinence. Dis Colon Rectum. 1996 Jan;39(1):59-65. doi: 10.1007/BF02048271. PMID 8601359
- [Background] Tan JJ, Chan M, Tjandra JJ. Evolving therapy for fecal incontinence. Dis Colon Rectum. 2007 Nov;50(11):1950-67. doi: 10.1007/s10350-007-9009-2. PMID 17874167
- [Background] Whitehead WE, Palsson OS, Simren M. Treating Fecal Incontinence: An Unmet Need in Primary Care Medicine. N C Med J. 2016 May-Jun;77(3):211-5. doi: 10.18043/ncm.77.3.211. PMID 27154893
- [Background] Zbar AP, Khaikin M. Should we care about the internal anal sphincter? Dis Colon Rectum. 2012 Jan;55(1):105-8. doi: 10.1097/DCR.0b013e318235b645. PMID 22156875
- [Background] Zutshi M, Tracey TH, Bast J, Halverson A, Na J. Ten-year outcome after anal sphincter repair for fecal incontinence. Dis Colon Rectum. 2009 Jun;52(6):1089-94. doi: 10.1007/DCR.0b013e3181a0a79c. PMID 19581851